CLINICAL TRIAL: NCT00758641
Title: Use of PRP to Treat Plantar Fasciitis, Blinded and Randomized as a Multi Center Study
Brief Title: Platelet Rich Plasma to Treat Plantar Fasciitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Elisabeth-TweeSteden Ziekenhuis (Other); Diaconessenhuis Leiden Netherlands (Unknown); Biomet Nederland BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BiometNL_16400076; Eudradact 2008-001257-18; CCMO 22305.008.08 BI
Record Dates: First submitted 2008-09-22; First posted 2008-09-25 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2016-06

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; platelet rich plasma; GPS
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- L-PRP Injection (Experimental): L-PRP produced with Biomet Recover L-PRP Platelet Separation Kit
  Interventions: Device: L-PRP Injection
- Steroid Injection (Active Comparator): Corticosteroid injections
  Interventions: Drug: Corticosteroid Injection

INTERVENTIONS:
Device: L-PRP Injection — L-PRP produced with Biomet Recover L-PRP Platelet Separation Kit
  Arms: L-PRP Injection
Drug: Corticosteroid Injection — kenacort 40 mg/ml triamcinolon acetonide
  Other Names: Corticosteroid
  Arms: Steroid Injection

SUMMARY:
Rationale: The standard treatment of chronic plantar fasciitis is corticosteroid injections. Corticosteroid injection give temporarily pain reduction, but no healing. Blood platelets initiate the natural healing rate. GPS ® gives an eightfold concentrate platelets of patients own blood. Injection of these platelets in the tendon might induce a healing rate.

Objective: To compare the efficacy of autologous platelet concentrate injections with corticosteroid injection in patients suffering from plantar fasciitis with respect to pain and function.

DETAILED DESCRIPTION:
Plantar fasciitis is the most common cause of foot complaints in the United States, making up 11 to 15 percent of the foot symptoms requiring professional care among adults (Pfeffer et al., 1999; Cole et al., 2005). A 2004 publication found that there are approximately 1 million patient visits per year to office-based physicians and hospital outpatient departments in the United States for plantar fasciitis (Riddle et al., 2004). This figure does not consider podiatric physicians visits, including these numbers would raise the overall physician visits related to plantar fasciitis considerably. The incidence of plantar fasciitis peaks in people between the ages of 40 to 60 years with no bias towards either sex (Taunton et al., 2002) The underlying condition that causes plantar fasciitis is a degenerative tissue condition that occurs near the site of origin of the plantar fascia at the medial tuberosity of the calcaneous (Buchbinder, 2004). In acute cases, plantar fasciitis is characterized by classical signs of inflammation including pain, swelling and loss of function. For more chronic conditions, however, inflammation is not the underlying tissue disruption. In fact, histology of chronic cases has shown no signs of inflammatory cell invasion into the affected area (Lemont et al., 2003). The tissue instead is characterized histological by infiltration with macrophages, lymphocytes, and plasma cells; tissue destruction; and repair involving immature vascularization and fibrosis (Lemont et al., 2003). The normal fascia tissue is replaced by an angiofibroblastic hyperplastic tissue which insuitates itself throughout the surrounding tissue creating a self-perpetuating cycle of degeneration (Lemont et al., 2003). In these chronic cases, the suffix 'itis' is a misnomer with plantar fasciosis being a more apt description of the underlying histology.

Conservative treatments including stretching protocols and foot orthoses resolve many cases of plantar fasciitis, with reports for patients in orthopedic practices being around 80 percent resolution (Cole et al., 2005; Wolgin et al., 1994; Martin et al., 1998; Davies et al., 1999). For more chronic cases, a number of non-surgical interventions are utilized including extracorperal shock wave therapy and corticosteroid injections (Cole et al., 2005; Speed et al., 2003; Acevedo, Beskin, 1998). The use of corticosteroids is particularly troubling as several studies have linked plantar fascial rupture to repeated local injections of a corticosteroid (Cole et al., 2005; Sellman, 1994; Leach et al., 1978; Acevedo, Beskin, 1998).

All of these methods are limited in their efficacy for cases of chronic plantar fasciitis due to the fact that none of them adequately addresses the full scope of the underlying tissue degeneration. This frequently leaves surgical intervention as the only viable option in these chronic cases.

The goal of treatment for chronic plantar fasciitis should be to cease and ultimately reverse the degenerating tissue disruption that is at the root of the condition. The three steps critical to full repair of the effected tissue are:

1. Enhancing the influx and proliferation of fibroblasts into the effected area. This will allow for a tissue bed that is extremely receptive to vascularization
2. Promote angiogenesis to develop a mature vascular structure in the effected area
3. With a mature vascularization, collagen deposition can then occur, resulting in the organization of fully mature tendon tissue

The injection of platelet-rich-plasma (PRP) into the effected tissue addresses all three healing stages necessary to reverse the degenerative process. The individual cytokines present in the platelet α-granules have been shown to enhance fibroblast migration and proliferation, upregulate vascularization, and increases collagen deposition in a variety of in vitro and in vivo settings [Molloy 2004]. Autologous PRP contains concentrated white blood cells and platelets that are suspended in plasma. Since an acidic anticoagulant (Anticoagulant Citrate Dextrose Solution A) is used to allow for processing of the whole blood via centrifugation, the PRP must be buffered to increase the pH to normal physiologic levels prior for injection into the effected tissue. This is accomplished with the addition of an 8.4% sodium bicarbonate solution at a ratio 0.05cc of sodium bicarbonate solution to 1cc of platelet concentrate. The resulting buffered platelet concentrate contains approximately 6 to 8 times concentration of platelets compared to baseline whole blood.

The cytokines present in platelet α-granules have been shown to affect the three healing stages necessary to reverse a chronic plantar fasciitis condition (Molloy et al., 2003). Additionally, many of these cytokines have been seen to work in a dose dependent manner (Molloy et al., 2003). A PRP injection into the effected area of tissue would provide concentrated levels of cytokines that should result in a healing cascade that halts and ultimately reverses the underlying pathology of elbow tendinosis. This treatment concept directly addresses the existing condition and should prove to be a superior alternative to current conservative treatments for chronic plantar fasciitis.

The objective of this clinical investigation is to compare the efficacy of autologous platelet concentrate injections with corticosteroid injection in patients suffering from plantar fasciitis with respect to pain and function.

Primary question Does injection with autologous platelet concentrate results in a larger percentage of successfully treated patients after 6 month as injection corticosteroid injection?

Secondary questions Does injection with autologous platelet concentrate has a larger pain reduction as injection of corticosteroid injection? (VAS) Does injection with autologous platelet concentrate has a larger improvement in function as corticosteroid injection? (AOFAS, WHOQol) Does injection with autologous platelet concentrate has a larger amount of satisfied patients as of corticosteroid injection? (WHOQol, satisfaction)

ELIGIBILITY:
Inclusion Criteria:

* No bias to sex
* > 18 years
* Chronic plantar fasciitis or proximal recalcitrant plantar heel pain (6-12 months duration)
* Failed conservative treatment
* Able to understand the informed consent
* VAS pain in morning by first steps higher as 5 (0-10 scale)

Exclusion Criteria:

* Received local steroid injections within 6 weeks, physical/occupational therapies within 4 weeks, or non-steroidal anti-inflammatory within 1 week prior to randomization
* Inability to fulfil follow-up criteria
* Significant cardiovascular, renal or hepatic disease
* Pregnant
* (Local) malignancy
* History of amenia (hemoglobin < 5.0 )
* Previous surgery for plantar fasciitis
* Active bilateral plantar fasciitis
* Diagnosis of vascular insufficiency or neuropathy related to heel pain
* Hypothyroidism
* Diabetics
* No other painful or function limited disorders of the foot and ankle

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-09; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Percentage of successfully treated patients | 6 months

SECONDARY OUTCOMES:
Pain reduction | 0-12 months
Function | 0-12 months
Patient satisfaction | 0-12 months
Complications and reinventions | 0-12 months

CONTACTS AND LOCATIONS:
Overall Officials: T Gosens, MD, PhD, Principal Investigator — St Elisabeth Hospital; H.M. Schuller, PhD, MD, Principal Investigator — Diaconessehuis Leiden
Locations (5):
- Netherlands (5):
  - Haga ziekenhuis, DenHaag
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Diaconessehuis, Leiden
  - Academisch Ziekenhuis Maastricht, Maastricht
  - St Elisabeth Hospital, Tilburg

REFERENCES:
- [Derived] Peerbooms JC, Lodder P, den Oudsten BL, Doorgeest K, Schuller HM, Gosens T. Positive Effect of Platelet-Rich Plasma on Pain in Plantar Fasciitis: A Double-Blind Multicenter Randomized Controlled Trial. Am J Sports Med. 2019 Nov;47(13):3238-3246. doi: 10.1177/0363546519877181. Epub 2019 Oct 11. PMID 31603721
- [Derived] Peerbooms JC, van Laar W, Faber F, Schuller HM, van der Hoeven H, Gosens T. Use of platelet rich plasma to treat plantar fasciitis: design of a multi centre randomized controlled trial. BMC Musculoskelet Disord. 2010 Apr 14;11:69. doi: 10.1186/1471-2474-11-69. PMID 20398269